CLINICAL TRIAL: NCT02023177
Title: Phase Angle as a Nutritional Marker Related to Prognosis Inpatients With Cirrhosis: A Cutt-off Value for Mexican Population
Brief Title: Phase Angle and Mortality in Patients With Cirrhosis
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Principal investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: PhA01
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Malnutrition
Keywords: phase angle; liver cirrhosis; mortality; malnutrition
MeSH Terms: conditions — Malnutrition; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Phase angle: Phase angle obtained from bioelectrical impedance

SUMMARY:
A few PhA cut-off points have been proposed to define malnutrition in cirrhosis, and they have proven to be useful in prognosticating severity of the disease and mortality. However, PhA needs specific validation in different ethnic groups. The aim of this study was to evaluate the PhA cut-off value that would best define malnutrition and predict mortality in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Malnutrition is a frequent complication of cirrhosis, and it has been associated with a more severe disease and decompensating events. Despite its relevance, there is no gold standard for nutritional assessment in cirrhosis, and intrinsic pathophysiologic changes make biochemical markers and traditional methods used to evaluate malnutrition unreliable. Phase angle (PhA) obtained from bioelectrical impedance has been successfully used as a nutritional marker in several diseases such as chronic renal failure, cancer, and HIV, where it has been associated with prolonged in-hospital stay and mortality. In cirrhosis, research linking malnutrition to increased mortality has yielded conflicting results, likely due to the lack of a gold standard. A few PhA cut-off points have been proposed to define malnutrition in cirrhosis, and they have proven to be useful in prognosticating severity of the disease and mortality. However, PhA needs specific validation in different ethnic groups. The aim of this study was to evaluate the PhA cut-off value that would best define malnutrition and predict mortality in patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old ambulatory patients Diagnosis of liver cirrhosis

Exclusion Criteria:

* Acute or chronic liver failure heart failure hepatocellular carcinoma pregnancy acute infections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be selected from the Liver Clinic at the Department of Gastroenterology in a tertiary care center in Mexico
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2008-01; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Baseline
  Phase angle obtained from bioelectrical impedance

OTHER OUTCOMES:
Nutritional status | 9 months
  Phase angle obtained from bioelectrical impedance
Nutritional status | 18 months
  Phase angle obtained from bioelectrical impedance
Nutritional status | 24 months
  Phase angle obtained from bioelectrical impedance

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, MD MSci, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Astrid Ruiz-Margáin, B.Sci, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico